CLINICAL TRIAL: NCT01889433
Title: An Open-label Randomized Multicenter Phase III Clinical Study Comparing Safety and Efficacy of Algeron (Cepeginterferon Alfa-2b) and Ribavirin With Pegasys (Peginterferon Alfa-2a) and Ribavirin for Treatment of Patients With Chronic Hepatitis C
Brief Title: An Open-label Comparative Efficacy and Safety Study of Algeron (Cepeginterferon Alfa-2b) in Treatment-naive Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCD-016-3
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Hepatitis; Hepatitis C
Keywords: Hepatitis C; Cepeginterferon alfa; Peginterferon; Treatment
MeSH Terms: conditions — Hepatitis; Hepatitis C | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Algeron (Experimental): Algeron at a dose of 1.5 µg/kg of body weight subcutaneously, once a week, and Rebetol, orally, at a daily dose of 800 mg (for body weight <65 kg), 1,000 mg (for body weight 65 - 85 kg), 1,200 mg (for body weight 86 - 105 kg) or 1,400 mg (for body weight > 105 kg).
  Interventions: Drug: Algeron
- Pegasys (Active Comparator): Pegasys in a dose of 180 µg subcutaneously, once a week, in combination with Rebetol, orally, at a daily dose of 800 mg for patients with genotype 2 or 3, and for genotypes 1 or 4 at a daily dose of 1000 mg (for body weight <75 kg) or 1200 mg (for body weight ≥75 kg)
  Interventions: Drug: Pegasys

INTERVENTIONS:
Drug: Algeron — 1.5 µg/kg of body weight subcutaneously, once a week
  Other Names: Cepeginterferon alfa-2b
  Arms: Algeron
Drug: Pegasys — 180 µg subcutaneously, once a week
  Other Names: Peginterferon alfa-2a
  Arms: Pegasys

SUMMARY:
The purpose of the study is to demonstrate the noninferiority of Algeron in combination with ribavirin compared to Pegasys in combination with ribavirin in the treatment of chronic hepatitis C.

DETAILED DESCRIPTION:
The course of treatment in both groups shall be 12 weeks, and efficacy analysis, i.e. rate of rapid (after the 4th week) and early (after the 12th week) virologic response will be based on PCR data. For patients with treatment failure after the 12th week the antiviral therapy shall be discontinued. All patients who require further anti-viral treatment will receive a combination treatment with Algeron / Pegasys and ribavirin for another 12 or 36 weeks (depending on the HCV genotype). Sustained virologic response will be assessed 24 weeks after last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Chronic HCV infection (genotypes 1а, 1b, 2, 3, 4) with detectable HCV RNA >6 month before the screening visit or abnormal ALT levels for >6 month before the screening visit.
3. Male and female patients, 18 to 70 years of age, inclusive.
4. Body mass index of 18 - 30 kg/m2.
5. Preserved protein synthetic liver function (INR < 1.7, albumin > 35 g/l).
6. No signs of hepatic encephalopathy or abdominal fluid retention according to clinical and ultrasound examination.
7. Fertile patients and their partners agree to use barrier contraception throughout the study treatment and 7 months after it.
8. Patient must have documentation of fibroscan within 1 year before the screening visit or agree to have a fibroscan within the screening period.

Exclusion Criteria:

1. Intolerance to IFN alfa, ribavirin or any components of this preparations confirmed by past medical history.
2. Infection by hepatitis B, A, E virus or HIV (co-infection).
3. Any other documented significant liver disease (drug or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, nonalcoholic steatohepatitis, biliary cirrohosis, etc.).
4. Past history of HCV treatment with IFN alfa or pegylated IFN alfa.
5. Administration of injectable and non-injectable interferons and/or some interferon inducers for any indication (other than HCV) for one month before enrollment into the study.
6. Cholestatic hepatitis (level of conjugated bilirubin, alkaline phosphatase, G-GTP exceeding the upper normal level by more than 5 times).
7. Decompensated liver cirrhosis confirmed by laboratory findings (class B, С according to Child-Pugh) or ultrasound examination.
8. Any documented autoimmune diseases (e.g., Crohn's disease, ulcerative colitis, systemic lupus erythematosus, idiopathic thrombocytopenic purpura, scleroderma, autoimmune haemolytic anemia, severe psoriasis).
9. Hemoglobin not lower than low normal level; neutrophils < 1.5 х109/L; platelets < 90 х109/L; creatinin level exceeding the upper normal level by more than 1.5 times, ALT level exceeding the upper normal level by more than 10 times.
10. Documented hemoglobinopathies (e.g., thalassemia major, sickle-cell anemia).
11. Severe depression, schizophrenia, other mental disorders, which from the investigator's point of view are a contraindication for anti-viral treatment.
12. Epilepsy and/or disorder of function of the central nervous system.
13. Abnormal thyroid function (TTH level beyond the normal values).
14. Diagnosed or suspected hepatocellular carcinoma as evidenced by screening alfa-fetoprotein (AFP) of ≥ upper normal level.
15. Antinuclear antibody (ANA) titer ≥1:640 at screening and/or evidence of autoimmune hepatitis on liver biopsy.
16. Malignant neoplasms.
17. Pregnancy, lactation period.
18. Severe comorbidities (for example, severe hypertension, severe coronary heart disease, decompensated diabetes mellitus) that represent a contraindication for anti-viral treatment.
19. Documented rare hereditary diseases, such as intolerance of lactose, sucrose, fructose, lactase deficiency or glucose-galactose malabsorption.
20. Known drug or alcohol abuse or signs of drug/alcohol abuse in present, which from the investigator's point of view are a contraindication for anti-viral treatment or restrict adherence to the treatment regimen.
21. Simultaneous participation in other clinical studies less than 30 days before enrollment into this study or previous participation in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
EVR | 12 weeks
  Proportion of randomized patients achieving early virologic response (EVR) - negative PCR result for HCV RNA (< 15 IU/ml) or ≥ 2log10 decrease of viral load after 12 weeks of study treatment

SECONDARY OUTCOMES:
RVR | 4 weeks
  Proportion of randomized patients achieving rapid virologic response (RVR) - negative PCR result for HCV RNA (< 15 IU/ml) after 4 weeks of treatment.
SVR (24) | 24 weeks after last dose of study treatment
  Proportion of randomized patients achieving sustained virologic response (SVR) - negative PCR result for HCV RNA (< 15 IU/ml) 24 weeks after last dose of study treatment
EOT | After 24 weeks of treatment for patients with genotype 2 or 3 and after 48 weeks of treatment for patients with genotype 1 or 4
  Proportion of randomized patients achieving end-of-treatment response (EOT) -undetectable HCV RNA (< 15 IU/ml) at the end of treatment (after 24 weeks of treatment for patients with genotype 2 or 3 and after 48 weeks of treatment for patients with genotype 1 or 4).
Biochemical Response | 12, 24, 48 weeks of treatment, and 24 weeks after last dose of study treatment
  Proportion of patients who have ALT level ≤ than upper normal level after 12 weeks of treatment, at the end of treatment (after 24 weeks of treatment for patients with genotype 2 or 3 and after 48 weeks of treatment for patients with genotype 1 or 4) and 24 weeks after last dose of study treatment.
Histological Response | 12 weeks of treatment and 24 weeks after last dose of study treatment
  Proportion of patients who have histological response, defined by a 1 level decrease in total METAVIR score measured on Fibroscan

OTHER OUTCOMES:
Immunogenicity | Week 0, 12, 24, and additionally for patients with HCV 1, 4 genotype - week 48 after first administration of Algeron / Pegasys and 24 weeks after last dose of study treatment
  Proportion of randomized patients with neutralizing antibodies to IFN alfa

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Zhdanov, Professor, Principal Investigator — Federal State Military Higher Vocational Education Institution S.M. Kirov Military Medical Academy; Olga Znoyko, Professor, Principal Investigator — State Budgetary Higher Vocational Education Institution A.I. Evdokimov Moscow State University of Medicine and Dentistry; Marina Maevskaya, Professor, Principal Investigator — State Budgetary Higher Vocational Education Institution I.M. Sechenov First Moscow State Medical University; Vjacheslav Morozov, Principal Investigator — LLC Medical Company "Hepatolog", Samara, Russia; Natalja Mironova, PhD, Principal Investigator — Municipal Healthcare Institution City Clinical Hospital No.2 named after V.I. Razumovsky, Healthcare Committee at the Administration of "Saratov City" Municipal District; Elena Nurmuhametova, PhD, Principal Investigator — State Public Healthcare Institution of the City of Moscow "Infectious Disease Clinical Hospital No. 1", Moscow City Health Department; Victor Pasechnikov, Professor, Principal Investigator — State Budgetary Higher Vocational Education Institution Stavropol State Medical Academy, Ministry of Health of the Russian Federation; Natalia Petrochenkova, PhD, Principal Investigator — State Budgetary Higher Vocational Education Institution Smolensk State Medical Academy; Tamara Sologub, Professor, Principal Investigator — Federal State Budgetary Institution Research Institute of Influenza, Ministry of Health of the Russian Federation, Saint-Petersburg; Vladimir Rafalskiy, Professor, Principal Investigator — Regional State Healthcare Institution "Smolensk Regional Clinical Hospital"; Evgeniy Chesnokov, Professor, Principal Investigator — State Medical and Preventive Institution of the Tyumen Region "Advisory and Diagnostic Center", Tyumen; Sandeep Gupta, Dr, Principal Investigator — M V Hospital & Research Center, 314/30 Mirza Mandi, Chowk 226003, Lucknow 226003, Uttar Pradesh, India; Tariq A Patil, Dr, Principal Investigator — Bhatia Hospital, Medical Research Society Tardeo Road, Grant Road (W), Maharashtra, India; Mandar Doiphode, Dr, Principal Investigator — Medipoint Hospitals Pvt. Ltd. Maharashtra, India; G S Malpani, Dr, Principal Investigator — Suyash Hospital Pvt. Ltd. Opposite M.G.M Medical College A.B. Road, Madhya Pradesh, India; Tawesak Tanwandee, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Faculty of Medicine, Siriraj Hospital, Bangkoknoi, Bangkok, Thailand; Thongsawat Satawat, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Faculty of Medicine, Chiang Mai University, Sriphum, Muang, Chiang Mai, Thailand
Locations (19):
- Belarus (2):
  - Gomel Regional Clinical Hospital, Homyel
  - Vitebsk Regional Clinical Hospital, Vitebsk
- India (4):
  - Suyash Hospital Pvt. Ltd. Opposite M.G.M Medical College A.B. Road, Indore
  - M V Hospital & Research Center, Lucknow
  - Bhatia Hospital, Medical Research Society Tardeo Road, Grant Road (W), Mumbai
  - Medipoint Hospitals Pvt. Ltd., Pune
- Russia (11):
  - State Budgetary Higher Vocational Education Institution A.I. Evdokimov Moscow State University of Medicine and Dentistry, Moscow
  - State Budgetary Higher Vocational Education Institution I.M. Sechenov First Moscow State Medical University, Moscow
  - State Public Healthcare Institution of the City of Moscow "Infectious Disease Clinical Hospital No. 1", Moscow
  - Federal State Budgetary Institution Research Institute of Influenza, Saint Petersburg
  - Federal State Military Higher Vocational Education Institution S.M. Kirov Military Medical Academy, Saint Petersburg
  - LLC Medical Company "Hepatolog", Samara
  - Municipal Healthcare Institution City Clinical Hospital No.2 named after V.I. Razumovsky, Saratov
  - Smolensk Regional Clinical Hospital, Smolensk
  - State Budgetary Higher Vocational Education Institution Smolensk State Medical Academy, Smolensk
  - State Budgetary Higher Vocational Education Institution Stavropol State Medical Academy, Stavropol
  - State Medical and Preventive Institution of the Tyumen Region "Advisory and Diagnostic Center", Tyumen
- Thailand (2):
  - Division of Gastroenterology, Department of Medicine, Faculty of Medicine, Siriraj Hospital, Bangkok
  - Division of Gastroenterology, Department of Internal Medicine, Faculty of Medicine, Chiang Mai University, Maharaj Nakorn Chiang Mai Hospital, Chiang Mai